CLINICAL TRIAL: NCT03348293
Title: Safety Study of 3D Printing Personalized Biodegradable Implant for Breast Reconstruction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20172047-1
Record Dates: First submitted 2017-09-15; First posted 2017-11-20 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: Breast Reconstruction; Breast Cancer
Keywords: biodegradable scaffold; immediate breast reconstruction; 3D printing
MeSH Terms: conditions — Breast Neoplasms | interventions — Printing, Three-Dimensional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3D printing patient (Experimental): Immediate breast reconstruction using 3D printing personalized scaffold
  Interventions: Procedure: 3D printing

INTERVENTIONS:
Procedure: 3D printing — Scope of tumor resection was simulated according to the MR imaging data. After meticulous design, we created the personalized porous biodegradable scaffold and printed by 3D printer, using porous PCL biomaterials. During operation, the biodegradable scaffold was implanted into the defective cavity after tumor resection.

SUMMARY:
Scope of tumor resection was simulated according to the MR imaging data. After meticulous design, the investigators created the personalized porous biodegradable scaffold and printed by 3D printer, using porous PCL biomaterials. During operation, the biodegradable scaffold was implanted into the defective cavity after tumor resection. Safety indicator, cosmetic outcome and autologous compatibility were evaluated.

DETAILED DESCRIPTION:
3D image reconstruction and printing Magnetic model images data were firstly produced by Siemens Trio Tim 3. 0 T MRI. The relative scanning parameters were adjusted as follows: layer thickness 0.9mm; pixel pitch 0.625 mm. In general, the thicker the layer thickness and pixel pitch, the better resolution and the more similar reconstructed model the investigators will get. The MRI data were then imported into Mimics 17.0® [Materialise, Leuven, Belgium] for 3D reconstruction of the targeted area. In this software, the investigators can adjust threshold value to acclimatize to segment tumor area. After that, 3D models were calculated and output as .stl files. According to the requirements of surgical planning, the scope of tumor resection was created after 2 cm expansion of the tumor area, that is, the filling scope of the implant. Next, the investigators designed the personalized porous degradable scaffold. In order to guarantee no significant differences and deformation of the implanted scaffold, the investigators used the contour of tumor resection as the boundary of the scaffold, with flexible porous structure as the units of the scaffold. Boolean operation can help to achieve this target. Finally, the printing of the personalized porous biodegradable scaffold was carried out. Biologically active material PCL was selected and the deformation and degradation time were set for 2 years by adjusting the molecular weight of PCL. Theoretically, PCL with the molecular weight above 65,000 can stably exist for 2 years in vivo, and then it will gradually degrade into H2O and CO2.The PCL material was put into the 3D printer, which was developed by the State key laboratory for mechanical manufacturing systems engineering of Xi'an Jiaotong university. The personalized porous biodegradable scaffold was completed after printing and removing supports.

Procedure In this study,the investigators produced the bio-implant at least 10 days before surgery. Before surgery, the printed bio-implant has been prepared and obtained full sterilization. Simply, under general anaesthesia, lumpectomy and sentinel-lymph-node biopsy was performed firstly, followed by 3D-printing scaffold transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients
* Tumor sized 3 cm to 6 cm
* ECOG score 1-2
* Multiple diffuse lesions in one quadrant
* Written informed consent

Exclusion Criteria:

* Triple negative breast cancer patients
* Participant in another clinical study
* Pregnancy and breastfeeding
* Patients with nipple infringement
* Inflammatory breast carcinoma
* Paget's disease
* Serious operative contraindication
* Contraindication for MRI

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
adverse events | 1 year after surgery
  Such adverse events include (but are not limited to) infection, repeated removal of implanted bio-scaffold, the humoral immunological responses.

SECONDARY OUTCOMES:
Cosmetic outcome | 6 months after surgery
  excellent (size and shape of reconstructed breast are identical to the original breast); good (deformity of the reconstructed breast involved less than 1/4 of the original breast; fair (deformity of the reconstructed breast involves less than 1/4-1/2 of the original breast); and poor (breast deformity involves more than 1/2 of the original breast).
Satisfaction of patients | 6 months after surgery
  The satisfaction of patients was investigated by self-made questionnaire
Recurrence rate | 5 year after surgery
  5 year recurrence was observed
5-Year disease free survival | 5 year after surgery
  5 year survival was observed

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chia HN, Wu BM. Recent advances in 3D printing of biomaterials. J Biol Eng. 2015 Mar 1;9:4. doi: 10.1186/s13036-015-0001-4. eCollection 2015. PMID 25866560
- [Background] Ibrahim AM, Jose RR, Rabie AN, Gerstle TL, Lee BT, Lin SJ. Three-dimensional Printing in Developing Countries. Plast Reconstr Surg Glob Open. 2015 Aug 10;3(7):e443. doi: 10.1097/GOX.0000000000000298. eCollection 2015 Jul. PMID 26301132
- [Background] The utility of 3D printing for surgical planning and patient-specific implant design for complex spinal pathologies: case report. J Neurosurg Spine. 2017 Apr;26(4):513-518. doi: 10.3171/2016.9.SPINE16371. Epub 2017 Jan 20. PMID 28106524